CLINICAL TRIAL: NCT06311097
Title: Dairy Products to Your Gut and Brain
Acronym: YourGutBrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other); APC Microbiome Ireland (Unknown)
Responsible Party: Principal Investigator, Henrik Munch Roager, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M402
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Constipation
Keywords: Diet; Fermented dairy; Gut-brain axis; Microbiota
MeSH Terms: conditions — Constipation | interventions — Cultured Milk Products

STUDY DESIGN:
Intervention Model Description: Two 4-week intervention periods separated by a washout period of at least 4 weeks.
  The crossover intervention will include 60 participants. Another 40 participants will only complete the first (baseline) visit.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented dairy (Experimental): The fermented dairy product is Arla A38® naturel 1,5% yogurt. The yogurt contains Lactobacillus acidophilus culture.
  Interventions: Other: Fermented dairy
- Non-fermented dairy (Placebo Comparator): The non-fermented dairy product is Arla® Letmælk 1,5% (semi-skimmed milk). The fermented- and non-fermented dairy products are isocaloric and matched in macronutrient content.
  Interventions: Other: Non-fermented dairy

INTERVENTIONS:
Other: Fermented dairy — Participants will consume 300g of yogurt daily for 4 weeks as an integral part of their habitual diet, substituting other food items.
  Arms: Fermented dairy
Other: Non-fermented dairy — Participants will consume 300g of milk daily for 4 weeks as an integral part of their habitual diet, substituting other food items.
  Arms: Non-fermented dairy

SUMMARY:
The goal of this intervention study is to compare the effects of fermented dairy and non-fermented dairy on bowel habits and cognitive performance in healthy women with defecations every other day or less. Furthermore, the study aims to explore underlying mechanisms linking the gut and the brain.

In addition, a sub-study will be conducted to explore differences in gut and brain measures between women with daily (reference group) and few (intervention group) weekly bowel movements, respectively, and to explore associations between measures of gut- and brain function.

DETAILED DESCRIPTION:
Participants in the intervention study (n=60) will consume 300g of fermented dairy (yogurt) or non-fermented dairy (milk) daily for 4 weeks. After a washout period of at least 4 weeks, the participants will consume the alternative dairy product (yogurt or milk) for 4 weeks. The participants will collect samples at home and be tested at the institute before and after each condition (yogurt or milk).

Participants in the sub-study (n=40) will not undergo any dairy interventions and they will only take part in the baseline assessments.

Prior to all visits at the institute, the participants are asked to complete some study activities at home, including:

* consumption of sweet corns to estimate whole gut transit time
* collection of fecal- and urine samples
* measurement of methane and hydrogen in breath
* reporting of gastrointestinal symptoms, including stool frequency and Bristol Stool Scale

During all visits at the institute, the participants will undergo tests and measurements, including:

* measurement of methane and hydrogen in fasting breath
* collection of fasting blood samples
* completion of cognitive tests
* recordings of electrophysiological signals of the gut and the brain
* completion of questionnaires assessing mood, quality of life, and physical activity, among others

ELIGIBILITY:
Inclusion Criteria:

* Self-reported defecations every second day or less (intervention study only)
* Willing to consume 300g milk/yogurt on a daily basis (intervention study only)
* Owns a smartphone (iOS 11.0 and later or Android 5.0 and up)
* Understand Danish or English

Exclusion Criteria:

* Current pregnancy or lactation
* Dairy allergy or intolerance
* Prior diagnosis of psychiatric or neurological illness
* Current diagnosis of depression, anxiety, or stress
* Prior diagnosis of metabolic or gastrointestinal disease (e.g., cardiovascular disease, diabetes, chronic constipation or diarrhea, inflammatory bowel diseases (IBD), celiac disease, small intestinal bacterial overgrowth (SIBO), cancer, etc.)
* Use of antibiotics within the last month
* Use of peroral corticosteroids (inhalers excepted)
* Use of medications that alter normal bowel function and metabolism (e.g., laxatives, antidiarrheal agents, narcotics, diuretics, anticonvulsants, etc.)
* Use of neuroactive medications (e.g., antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinsonian, etc.)
* Concurrent participation in another trial
* Any condition that makes the project responsible researcher doubt the feasibility of the volunteer´s participation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline in defecation frequency between the interventions | Baseline and 4 weeks
  Participants will report all bowel movements in a defecation diary in the week leading up to the intervention (baseline) and in the last week of the intervention (week 4)

SECONDARY OUTCOMES:
Difference in change from baseline in cognitive performance between the interventions | Baseline and 4 weeks
  Changes in cognitive performance will be quantified by cognitive index comprising memory, attention, and psychomotor speed. A composite cognitive score will be calculated as the standard score. Z-score will be assessed with the baseline variance between 0 and 1. Memory: number of errors made by the participant. Lower number of errors indicating better outcome. Attention: latency (speed of response), probability of false alarms and sensitivity. Faster speed of response indicating better outcome and lower number of false alarms indicating better outcome. Psychomotor speed: lower values indicating faster reaction time and better outcome
Difference in change from baseline in phase-amplitude coupling between gastric slow-wave activity and cortical alpha activity between the interventions | Baseline and 4 weeks
  Gastric and cortical electrical activity will be measured by electrogastrography (EGG) and electroencephalography (EEG), respectively, to investigate the phase-amplitude coupling between the infra-slow (~ 0.05 Hz) gastric phase and the amplitude of the cortical alpha rhythm (10-11 Hz)
Difference in change from baseline in whole gut transit time between the interventions | Baseline and 4 weeks
  Whole gut transit time will be estimated by sweet-corn passage time
Difference in change from baseline in stool consistency between the interventions | Baseline and 4 weeks
  Changes in stool consistency will be estimated by the Bristol Stool Scale. The scale ranges from type 1 (hard stool) to type 7 (loose stool)
Difference in change from baseline in stool moisture between the interventions | Baseline and 4 weeks
  Fecal water content in percentage of stool weight will be measured
Difference in change from baseline in fecal abundance of Lactobacillus acidophilus between the interventions | Baseline and 4 weeks
  Marker of compliance. Will be assessed by fecal microbiota sequencing
Difference in change from baseline in self-reported gastrointestinal symptoms between the interventions | Baseline and 4 weeks
  Changes in subjective gastrointestinal symptoms will be reported by participants using a visual analog scale.The scale ranges from 0 (no symptoms) to 10 (very bad symptoms)

OTHER OUTCOMES:
Difference in change from baseline in gut microbiota between the interventions | Baseline and 4 weeks
  Fecal samples will be utilized for microbiota analyses (e.g., shotgun metagenome sequencing, 16S rRNA gene sequencing, and real-time PCR of selected bacterial taxa)
Difference in change from baseline in fecal pH between the interventions | Baseline and 4 weeks
  pH will be measured in fecal samples
Difference in change from baseline in breath hydrogen and methane levels between the interventions | Baseline and 4 weeks
  Changes in fasting breath hydrogen and methane concentrations will be measured in parts per million (PPM) in exhalations.Furthermore, breath hydrogen and methane concentrations will be measured (in PPM), twice daily (morning and evening) during each 4 week intervention using a portable breath analyzer
Difference in change from baseline in biomarkers of colonic fermentation between the interventions | Baseline and 4 weeks
  Fecal samples will be used for measurements of biomarkers of colonic fermentation. These markers include fecal nitrogen to carbon ratio, fecal ammonia, fecal redox potential, fecal energy density, fecal calprotectin, fecal proteolytic and saccharolytic enzymatic activity
Difference in change from baseline in fecal short-chain fatty acids (SCFAs) between the interventions | Baseline and 4 weeks
  Fecal concentrations of SCFAs will be quantified using mass spectrometry
Difference in change from baseline in fecal zonulin levels between the interventions | Baseline and 4 weeks
  Fecal zonulin levels will be measured via fecal samples
Difference in change from baseline in plasma levels of lipopolysaccharide-binding protein (LBP) between the interventions | Baseline and 4 weeks
  Plasma levels of LBP, a biomarker of intestinal permeability, will be measured by ELISA (enzyme-linked immunosorbent assay)
Difference in change from baseline in gut metabolome between the interventions | Baseline and 4 weeks
  Gut (fecal) metabolomes will be assessed by metabolomics
Difference in change from baseline in urine metabolome between the interventions | Baseline and 4 weeks
  Urine metabolomes will be assessed by untargeted metabolomics
Difference in change from baseline in plasma metabolome between the interventions | Baseline and 4 weeks
  Plasma metabolomes will be assessed by metabolomics
Difference in change from baseline in inflammatory biomarkers between the interventions | Baseline and 4 weeks
  The following inflammatory biomarkers will be measured in fasting blood samples: soluble urokinase plasminogen activator receptor (suPAR), C-reactive protein (CRP), interleukin 6 (IL-6) and tumor necrosis factor alpha (TNFα)
Difference in change from baseline in plasma levels of cortisol between the interventions | Baseline and 4 weeks
  Plasma cortisol levels will be measured in fasting blood samples
Difference in change from baseline in biomarkers of glucose and lipid metabolism between the interventions | Baseline and 4 weeks
  The following biomarkers of glucose and lipid metabolism will be measured in fasting blood samples: glucose, insulin, glucagon, total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides
Difference in change from baseline in appetite hormones between the interventions | Baseline and 4 weeks
  The following appetite hormones will be measured in fasting blood samples: glucagon-like peptide-1 (GLP-1), peptide YY (PYY), glucose-dependent insulinotropic polypeptide (GIP) and cholecystokinin (CCK)
Difference in change from baseline in plasma level of Brain Derived Neurotrophic Factor (BDNF) between the interventions | Baseline and 4 weeks
  Plasma levels of BDNF will be measured by ELISA
Difference in change from baseline in self-reported stress and mood between the interventions | Baseline and 4 weeks
  Self-reported stress and mood will be assessed by a 42 item scale that measures negative emotional states of depression, anxiety and stress (DASS-42). The scale ranges from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time)
Difference in change from baseline in self-reported sleeping patterns between the interventions | Baseline and 4 weeks
  Sleep pattern and quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI) at all visits. The PSQI consists of 19 items, summed into seven component scores and one overall composite score. Each item is rated on a scale from 0-3 with lower scores reflecting healthier sleep quality
Difference in change from baseline in resting-state cortical connectivity between the interventions | Baseline and 4 weeks
  Resting-state cortical connectivity will be measured using EEG during a period of rest at all visits
Difference in change from baseline in event-related potentials evoked by a cognitive task between the interventions | Baseline and 4 weeks
  Event-related potentials evoked by a cognitive task will be measured using EEG during a period of rest at all visits
Difference in change from baseline in quality of life between the interventions | Baseline and 4 weeks
  Quality of life will be assessed by the 36-Item short form survey (SF-36) at all visits. A score ranging from 0 to 100 will be obtained. Higher scores indicate better quality of life
Difference in change from baseline in habitual diet between the interventions | Baseline and 4 weeks
  Participants will record their food intake via MyFood24 for 3 days (one weekend day and two workdays) prior to all visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark